CLINICAL TRIAL: NCT02656290
Title: Prospective, Non-Randomized, Single Arm, Multicenter Clinical Evaluation of the Edwards Pericardial Aortic Bioprosthesis (Model 11000A) for Pulmonary Valve Replacement
Brief Title: COMMENCE Pulmonary: Clinical Evaluation of Edwards Pericardial Aortic Bioprosthesis (Model 11000A) for Pulmonary Valve Replacement
Acronym: COMMENCE-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-03
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Valve Insufficiency; Pulmonary Valve Degeneration; Congenital Pulmonary Valve Abnormality
MeSH Terms: conditions — Pulmonary Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Edwards Pericardial Aortic Bioprosthesis Model 11000A (Experimental): Pulmonary valve replacement
  Interventions: Device: Edwards Pericardial Aortic Bioprosthesis Model 11000A

INTERVENTIONS:
Device: Edwards Pericardial Aortic Bioprosthesis Model 11000A — Edwards Aortic Bioprosthesis Model 11000A in the pulmonary position; a trileaflet bioprosthesis comprised of bovine pericardium

SUMMARY:
The objective of this trial is to assess the safety and effectiveness of the Edwards Pericardial Aortic Bioprosthesis Model 11000A, in the pulmonary position in pediatric and adult subjects five years or older requiring replacement of their native or prosthetic pulmonary valve.

DETAILED DESCRIPTION:
This is a prospective, Non-Randomized, Single Arm, Multicenter study. Up to one hundred (100) pulmonary valve replacement (PVR) subjects at up to ten (10) clinical sites will be enrolled. Clinical data will be collected from at least 3 centers with data available on patients who have completed the 1 year follow-up visit. Subjects will be followed for and assessed after implant for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Has pulmonary valve disease requiring pulmonary valve replacement of their native or prosthetic valve
2. Is greater than or equal to 5 years of age
3. Subject and/or subject's legal representative has provided written informed consent as approved and required by the respective institutional review board and agrees to its provisions. NOTE: Written consent must be obtained prior to any research related test being performed.

Exclusion criteria:

A subject meeting any of the following criteria shall be excluded:

1. Valve-in-conduit procedure
2. Requires emergency surgery
3. Has acute myocardial infarction (MI) within 30 days prior to screening date
4. Has MRI or CT scan confirmed stroke, cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months (180 days) prior to screening date
5. Has hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 30 days prior to screening date
6. Has active endocarditis/myocarditis or endocarditis/myocarditis within 3 months prior to screening date
7. Has renal insufficiency as determined by creatinine (S-Cr) level ~ 2.5 mg/dL within 60 days prior to screening visit or end-stage renal disease
8. Has documented leukopenia (WBC < 3.5x 103/I-lL), acute anemia (Hgb <10.0 g/dL or 6 mmol/L), or thrombocytopenia (platelet count < 50xl03/I-lL) accompanied by history of bleeding diathesis or coagulopathy within 60 days prior to screening date
9. Diagnosed with abnormal calcium metabolism and/or hyperparathyroidism
10. Echocardiographic evidence of an intra-cardiac mass, thrombus, or vegetation
11. RVOT aneurysm unless treated during pulmonary valve replacement surgery
12. Has prior organ transplant or is currently an organ transplant candidate
13. Was previously implanted with INSPIRIS RESILIA Pulmonary valve
14. Previously implanted with an aortic, mitral, or tricuspid bioprosthetic valve, mechanical valve, or annuloplasty ring
15. Need for concomitant replacement of the aortic, mitral or tricuspid valves
16. Has presence of non-cardiac disease limiting life expectancy to less than 12 months
17. Is Currently or has recently participated (within 6 weeks) in another investigational drug or device trial
18. Positive urine or serum pregnancy test in female subjects of child-bearing potential and/or nursing mothers, or planning to become pregnant within 1 year of study valve implant
19. Has left ventricular ejection fraction ≤20% as validated by diagnostic procedure prior to screening date
20. Currently incarcerated or unable to give voluntary informed consent
21. Documented history of substance (drug or alcohol) abuse within the last 5 years prior to screening date
22. Patients with hypersensitivity to metal alloys that contain cobalt, chromium, nickel, molybdenum, manganese, carbon, beryllium and iron
23. Patients with hypersensitivity to latex

    Intra-Op Exclusion Criterion:
24. Significant injury to the heart upon entry defined as emergent cardiopulmonary bypass requiring femoral cannulation

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Baird, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers

RESULTS

PARTICIPANT FLOW:
Groups:
- Edwards Pericardial Aortic Bioprosthesis Model 11000A: Edwards Pericardial Aortic Bioprosthesis Model 11000A in the pulmonary position in subjects five years or older requiring replacement of their native or prosthetic pulmonary valve.
Period: Overall Study
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Started | 26
Discharge | 26
30 Days | 26
3-6 Months | 25
1 Year | 25
2 Years | 24
3 Years | 24
4 Years | 19
5 Years | 22
Completed | 22
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Reintervention | 3

BASELINE CHARACTERISTICS:
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subject's With Freedom From Device or Procedure Related Death and/or Reoperation at 1-year Post-implant.
Description: Subject's freedom from device or procedure related death and/or reoperation at 1-year post-implant. Time to events were estimated by Kaplan-Meier method. A higher number means a better outcome.
Time Frame: 1-year post-implant
Population: The outcome is reported for subjects who received the Edwards Pericardial Aortic Bioprosthesis Model 11000A device in the pulmonary position where data is available.
Measure: Number; unit: percentage of subjects
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 26
percentage of subjects | 100.0

2. Secondary Outcome: Percentage of Early Adverse Events
Description: Number of early adverse events occurring within 30 days of procedure divided by the total number of enrolled subjects times 100.
Time Frame: Percentage of events occurring within 30 days of procedure
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 26
percentage of subjects
  All Cause Death | 0.0
  Valve Related Death | 0.0
  All Paravalvular Leak (PVL) | 0.0
  All Transvalvular Leak (TVL) | 0.0
  Major Transvalvular Leak | 0.0
  Minor Transvalvular Leak | 0.0
  Endocarditis | 0.0
  Reintervention | 0.0
  Explant | 0.0
  Thromboembolism | 0.0
  Structural Valve Deterioration | 0.0
  Non-Structural Valve Deterioration Other than Paravalvular Leak | 0.0
  Valve Thrombosis - Pulmonary | 0.0
  All Bleeding | 3.8
  Major Bleeding | 3.8
  Minor Bleeding | 0.0
  Hemolysis | 0.0

3. Secondary Outcome: Number of Late Adverse Events Divided by Late Patient Years (Expressed as a Percentage) for the Trial Valve Cohort.
Description: Late patient years are calculated from 31 days post-implant to the date of the last follow-up visit (or contact) or adverse event. Late patient year calculation: [(Number of late events/sum of late patient years) x 100]
Time Frame: Events occurring ≥ 31 days and up through 5 years post implant.
Population: The outcome is reported for subjects who received the Edwards Pericardial Aortic Bioprosthesis Model 11000A in the pulmonary position where data is available.
Measure: Number; unit: Percentage of events/late patient years
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 26
Percentage of events/late patient years
  All cause death | 0.0
  Valve related death | 0.0
  All Paravalvular leak (PVL) | 0.0
  All Transvalvular Leak (TVL) | 13.7
  Major Transvalvular Leak | 2.3
  Minor Transvalvular | 11.4
  Endocarditis | 0.0
  Reintervention | 2.3
  Explant | 0.0
  Thromboembolism | 0.0
  Structural Valve Deterioration | 2.3
  Non-Structural Valve Deterioration other than PVL | 0.0
  Valve Thrombosis - Pulmonary | 0.0
  All Bleeding | 0.8
  Major Bleeding | 0.0
  Minor Bleeding | 0.8
  Hemolysis | 0.0

4. Secondary Outcome: Subject's Average Mean Gradient Measurements Over Time.
Description: Mean gradient is the average flow of blood through the aortic valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. In general, a higher value is considered worse, and a lower value is considered better but the value is dependent on the size and type of valve.
Time Frame: Baseline, 30 days, 3 months, and annually thereafter for up to 5 years
Population: This outcome is reported for subjects who received the trial valve. Note that the number of participants analyzed is different from that in the participant flow as there was some missing data.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Edwards Pericardial Aortic Bioprosthesis Model 11000A - 21 mm; Edwards Pericardial Aortic Bioprosthesis Model 11000A - 23 mm; Edwards Pericardial Aortic Bioprosthesis Model 11000A - 25 mm; Edwards Pericardial Aortic Bioprosthesis Model 11000A - 27 mm: Edwards Pericardial Aortic Bioprosthesis Model 11000A in the pulmonary position in subjects five years or older requiring replacement of their native or prosthetic pulmonary valve.
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 21 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 23 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 25 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 27 mm
Number analyzed (Participants) | 1 | 3 | 12 | 10
mmHg
  Baseline: number analyzed (Participants) | 0 | 3 | 9 | 7
  Baseline |  | 8.0 (1.7) | 9.0 (8.6) | 8.4 (3.0)
  30 days: number analyzed (Participants) | 0 | 0 | 8 | 7
  30 days |  |  | 7.7 (2.5) | 7.8 (2.8)
  3 months: number analyzed (Participants) | 1 | 2 | 10 | 6
  3 months | 9.5 (NA) — The sample size is 1 and therefore no standard deviation is available. | 12.9 (3.5) | 9.5 (3.3) | 8.8 (2.1)
  1 Year: number analyzed (Participants) | 1 | 0 | 10 | 9
  1 Year | 15.0 (NA) — The sample size is 1 and therefore no standard deviation is available. |  | 10.9 (4.3) | 10.3 (4.2)
  2 Years: number analyzed (Participants) | 1 | 1 | 10 | 7
  2 Years | 14.4 (NA) — The sample size is 1 and therefore no standard deviation is available. | 14.3 (NA) — The sample size is 1 and therefore no standard deviation is available. | 10.8 (3.8) | 10.7 (3.7)
  3 Years: number analyzed (Participants) | 1 | 1 | 10 | 9
  3 Years | 35.1 (NA) — The sample size is 1 and therefore no standard deviation is available. | 24.9 (NA) — The sample size is 1 and therefore no standard deviation is available. | 10.8 (3.5) | 11.7 (5.1)
  4 Years: number analyzed (Participants) | 0 | 0 | 9 | 5
  4 Years |  |  | 11.4 (3.1) | 11.3 (4.3)
  5 Years: number analyzed (Participants) | 1 | 0 | 7 | 8
  5 Years | 44.6 (NA) — The sample size is 1 and therefore no standard deviation is available. |  | 11.8 (2.6) | 10.9 (4.4)

5. Secondary Outcome: Subject's Average Peak Gradient Measurements Over Time.
Description: Peak gradient is the maximum value measured of flow of blood through the aortic valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. In general, a higher value is considered worse, and a lower value is considered better but the value is dependent on the size and type of valve.
Time Frame: Baseline, 30 days, 3 months, and annually thereafter for up to 5 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 21 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 23 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 25 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 27 mm
Number analyzed (Participants) | 1 | 3 | 12 | 10
mmHg
  Baseline: number analyzed (Participants) | 0 | 3 | 9 | 7
  Baseline |  | 15.6 (2.9) | 16.1 (14.4) | 16.4 (5.5)
  30 days: number analyzed (Participants) | 0 | 0 | 8 | 7
  30 days |  |  | 13.7 (4.5) | 13.6 (4.8)
  3 months: number analyzed (Participants) | 1 | 2 | 10 | 6
  3 months | 17.0 (NA) — The sample size is 1 and therefore no standard deviation is available. | 22.5 (5.3) | 16.7 (6.2) | 15.5 (3.2)
  1 Year: number analyzed (Participants) | 1 | 0 | 10 | 9
  1 Year | 26.8 (NA) — The sample size is 1 and therefore no standard deviation is available. |  | 19.1 (7.4) | 18.3 (7.5)
  2 Years: number analyzed (Participants) | 1 | 1 | 10 | 7
  2 Years | 23.4 (NA) — The sample size is 1 and therefore no standard deviation is available. | 23.8 (NA) — The sample size is 1 and therefore no standard deviation is available. | 19.4 (6.7) | 19.1 (6.4)
  3 Years: number analyzed (Participants) | 1 | 1 | 10 | 9
  3 Years | 62.4 (NA) — The sample size is 1 and therefore no standard deviation is available. | 42.0 (NA) — The sample size is 1 and therefore no standard deviation is available. | 19.2 (6.5) | 20.6 (8.9)
  4 Years: number analyzed (Participants) | 0 | 0 | 9 | 5
  4 Years |  |  | 19.9 (5.0) | 19.7 (7.3)
  5 Years: number analyzed (Participants) | 1 | 0 | 7 | 8
  5 Years | 77.8 (NA) — The sample size is 1 and therefore no standard deviation is available. |  | 20.9 (5.0) | 19.8 (7.9)

6. Secondary Outcome: Amount of Paravalvular Pulmonary Regurgitation in Subjects Over Time by Valve Size
Description: Paravalvular leak refers to blood flowing through a channel between the implanted artificial valve and the cardiac tissue as a result of inappropriate sealing. Paravalvular leak is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation/leak (a better outcome) and 4 represents severe regurgitation/leak (a worse outcome).
Time Frame: Discharge, 30 days, 3 months, and annually thereafter for up to 5 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 21 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 23 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 25 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 27 mm
Number analyzed (Participants) | 1 | 3 | 12 | 10
Participants
  Discharge: number analyzed (Participants) | 1 | 3 | 11 | 10
  Discharge: None (0) | 1 | 3 | 8 | 10
  Discharge: Trival/Trace (+1) | 0 | 0 | 3 | 0
  Discharge: Mild (+2) | 0 | 0 | 0 | 0
  Discharge: Moderate (+3) | 0 | 0 | 0 | 0
  Discharge: Severe (+4) | 0 | 0 | 0 | 0
  30 days: number analyzed (Participants) | 0 | 1 | 10 | 8
  30 days: None (0) |  | 1 | 9 | 8
  30 days: Trival/Trace (+1) |  | 0 | 1 | 0
  30 days: Mild (+2) |  | 0 | 0 | 0
  30 days: Moderate (+3) |  | 0 | 0 | 0
  30 days: Severe (+4) |  | 0 | 0 | 0
  3 months: number analyzed (Participants) | 1 | 3 | 11 | 7
  3 months: None (0) | 1 | 3 | 11 | 7
  3 months: Trival/Trace (+1) | 0 | 0 | 0 | 0
  3 months: Mild (+2) | 0 | 0 | 0 | 0
  3 months: Moderate (+3) | 0 | 0 | 0 | 0
  3 months: Severe (+4) | 0 | 0 | 0 | 0
  1 year: number analyzed (Participants) | 1 | 2 | 11 | 9
  1 year: None (0) | 1 | 2 | 10 | 9
  1 year: Trival/Trace (+1) | 0 | 0 | 1 | 0
  1 year: Mild (+2) | 0 | 0 | 0 | 0
  1 year: Moderate (+3) | 0 | 0 | 0 | 0
  1 year: Severe (+4) | 0 | 0 | 0 | 0
  2 years: number analyzed (Participants) | 1 | 2 | 11 | 8
  2 years: None (0) | 1 | 2 | 11 | 7
  2 years: Trival/Trace (+1) | 0 | 0 | 0 | 1
  2 years: Mild (+2) | 0 | 0 | 0 | 0
  2 years: Moderate (+3) | 0 | 0 | 0 | 0
  2 years: Severe (+4) | 0 | 0 | 0 | 0
  3 years: number analyzed (Participants) | 1 | 2 | 10 | 9
  3 years: None (0) | 1 | 2 | 10 | 9
  3 years: Trival/Trace (+1) | 0 | 0 | 0 | 0
  3 years: Mild (+2) | 0 | 0 | 0 | 0
  3 years: Moderate (+3) | 0 | 0 | 0 | 0
  3 years: Severe (+4) | 0 | 0 | 0 | 0
  4 years: number analyzed (Participants) | 0 | 1 | 10 | 5
  4 years: None (0) |  | 1 | 10 | 5
  4 years: Trival/Trace (+1) |  | 0 | 0 | 0
  4 years: Mild (+2) |  | 0 | 0 | 0
  4 years: Moderate (+3) |  | 0 | 0 | 0
  4 years: Severe (+4) |  | 0 | 0 | 0
  5 years: number analyzed (Participants) | 1 | 1 | 8 | 8
  5 years: None (0) | 1 | 1 | 8 | 8
  5 years: Trival/Trace (+1) | 0 | 0 | 0 | 0
  5 years: Mild (+2) | 0 | 0 | 0 | 0
  5 years: Moderate (+3) | 0 | 0 | 0 | 0
  5 years: Severe (+4) | 0 | 0 | 0 | 0

7. Secondary Outcome: Amount of Transvalvular Pulmonary Regurgitation in Subjects Over Time by Valve Size
Description: Valvular regurgitation occurs when the valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation (a better outcome) and 4 represents severe regurgitation (a worse outcome).
Time Frame: Discharge, 30 days, 3 months, and annually thereafter for up to 5 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 21 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 23 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 25 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 27 mm
Number analyzed (Participants) | 1 | 3 | 12 | 10
Participants
  Discharge: number analyzed (Participants) | 1 | 3 | 11 | 10
  Discharge: None (0) | 0 | 0 | 0 | 0
  Discharge: Trival/Trace (+1) | 1 | 3 | 11 | 9
  Discharge: Mild (+2) | 0 | 0 | 0 | 1
  Discharge: Moderate (+3) | 0 | 0 | 0 | 0
  Discharge: Severe (+4) | 0 | 0 | 0 | 0
  30 days: number analyzed (Participants) | 0 | 1 | 10 | 8
  30 days: None (0) |  | 0 | 0 | 0
  30 days: Trival/Trace (+1) |  | 1 | 10 | 6
  30 days: Mild (+2) |  | 0 | 0 | 2
  30 days: Moderate (+3) |  | 0 | 0 | 0
  30 days: Severe (+4) |  | 0 | 0 | 0
  3 months: number analyzed (Participants) | 1 | 3 | 11 | 7
  3 months: None (0) | 0 | 0 | 3 | 0
  3 months: Trival/Trace (+1) | 0 | 1 | 7 | 6
  3 months: Mild (+2) | 1 | 2 | 1 | 1
  3 months: Moderate (+3) | 0 | 0 | 0 | 0
  3 months: Severe (+4) | 0 | 0 | 0 | 0
  1 year: number analyzed (Participants) | 1 | 2 | 11 | 10
  1 year: None (0) | 0 | 0 | 1 | 0
  1 year: Trival/Trace (+1) | 0 | 0 | 7 | 5
  1 year: Mild (+2) | 1 | 2 | 2 | 3
  1 year: Moderate (+3) | 0 | 0 | 1 | 0
  1 year: Severe (+4) | 0 | 0 | 0 | 2
  2 years: number analyzed (Participants) | 1 | 2 | 11 | 8
  2 years: None (0) | 0 | 0 | 0 | 0
  2 years: Trival/Trace (+1) | 0 | 0 | 6 | 2
  2 years: Mild (+2) | 1 | 1 | 2 | 5
  2 years: Moderate (+3) | 0 | 1 | 3 | 0
  2 years: Severe (+4) | 0 | 0 | 0 | 1
  3 years: number analyzed (Participants) | 1 | 2 | 10 | 9
  3 years: None (0) | 0 | 0 | 0 | 0
  3 years: Trival/Trace (+1) | 0 | 0 | 4 | 3
  3 years: Mild (+2) | 0 | 1 | 2 | 3
  3 years: Moderate (+3) | 1 | 0 | 3 | 2
  3 years: Severe (+4) | 0 | 1 | 1 | 1
  4 years: number analyzed (Participants) | 0 | 1 | 10 | 5
  4 years: None (0) |  | 0 | 0 | 0
  4 years: Trival/Trace (+1) |  | 0 | 2 | 1
  4 years: Mild (+2) |  | 0 | 3 | 1
  4 years: Moderate (+3) |  | 0 | 3 | 2
  4 years: Severe (+4) |  | 1 | 2 | 1
  5 years: number analyzed (Participants) | 1 | 1 | 8 | 8
  5 years: None (0) | 0 | 0 | 0 | 0
  5 years: Trival/Trace (+1) | 0 | 0 | 1 | 2
  5 years: Mild (+2) | 0 | 0 | 2 | 0
  5 years: Moderate (+3) | 0 | 0 | 4 | 3
  5 years: Severe (+4) | 1 | 1 | 1 | 3

8. Secondary Outcome: Subject's Average Tricuspid Regurgitation (TR) Gradient Measurement Over Time.
Description: Tricuspid regurgitation (TR) gradient (peak systolic) is defined as the maximum value measured of blood flowing back through the tricuspid valve during systole as measured in millimeters of mercury. In general, a higher value is considered worse, and a lower value is considered better but the value is dependent on the size and type of valve.
Time Frame: Baseline, 30 days, 3 months, and annually thereafter for up to 5 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 21 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 23 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 25 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 27 mm
Number analyzed (Participants) | 1 | 3 | 12 | 10
mmHg
  Baseline: number analyzed (Participants) | 0 | 2 | 8 | 5
  Baseline |  | 21.5 (0.6) | 36.2 (30.6) | 28.8 (6.1)
  30 days: number analyzed (Participants) | 0 | 0 | 7 | 6
  30 days |  |  | 30.8 (9.3) | 25.2 (7.2)
  3 months: number analyzed (Participants) | 0 | 2 | 8 | 6
  3 months |  | 31.6 (7.3) | 32.9 (9.4) | 28.8 (6.9)
  1 Year: number analyzed (Participants) | 1 | 1 | 9 | 8
  1 Year | 23.6 (NA) — The sample size is 1 and therefore no standard deviation is available. | 30.2 (NA) — The sample size is 1 and therefore no standard deviation is available. | 27.7 (7.4) | 27.7 (3.8)
  2 Years: number analyzed (Participants) | 0 | 1 | 8 | 7
  2 Years |  | 27.7 (NA) — The sample size is 1 and therefore no standard deviation is available. | 30.9 (9.7) | 24.0 (8.0)
  3 Years: number analyzed (Participants) | 0 | 1 | 9 | 7
  3 Years |  | 37.2 (NA) — The sample size is 1 and therefore no standard deviation is available. | 29.2 (12.0) | 29.2 (7.7)
  4 Years: number analyzed (Participants) | 0 | 1 | 7 | 5
  4 Years |  | 28.0 (NA) — The sample size is 1 and therefore no standard deviation is available. | 35.5 (8.9) | 29.9 (10.1)
  5 Years: number analyzed (Participants) | 0 | 1 | 7 | 7
  5 Years |  | 42.8 (NA) — The sample size is 1 and therefore no standard deviation is available. | 30.3 (8.5) | 29.4 (8.3)

9. Secondary Outcome: Subject's Average Peak Velocity Measurement Over Time
Description: Peak velocity is defined as the maximum speed in meters per second that the blood is flowing through the pulmonic heart valve in a given direction. In general, a higher value is considered worse, and a lower value is considered better but the value is dependent on the size and type of valve.
Time Frame: Baseline, 30 days, 3 months, and annually thereafter for up to 5 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 21 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 23 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 25 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 27 mm
Number analyzed (Participants) | 1 | 3 | 12 | 10
m/s
  Baseline: number analyzed (Participants) | 0 | 3 | 9 | 7
  Baseline |  | 2.0 (0.2) | 1.8 (0.8) | 2.0 (0.4)
  30 days: number analyzed (Participants) | 0 | 0 | 8 | 7
  30 days |  |  | 1.8 (0.3) | 1.8 (0.3)
  3 Months: number analyzed (Participants) | 1 | 2 | 10 | 6
  3 Months | 2.1 (NA) — The sample size is 1 and therefore no standard deviation is available. | 2.4 (0.3) | 2.0 (0.4) | 2.0 (0.2)
  1 Year: number analyzed (Participants) | 1 | 0 | 10 | 9
  1 Year | 2.6 (NA) — The sample size is 1 and therefore no standard deviation is available. |  | 2.2 (0.4) | 2.1 (0.4)
  2 Years: number analyzed (Participants) | 1 | 1 | 10 | 7
  2 Years | 2.4 (NA) — The sample size is 1 and therefore no standard deviation is available. | 2.4 (NA) — The sample size is 1 and therefore no standard deviation is available. | 2.2 (0.4) | 2.2 (0.4)
  3 Years: number analyzed (Participants) | 1 | 1 | 10 | 9
  3 Years | 4.0 (NA) — The sample size is 1 and therefore no standard deviation is available. | 3.2 (NA) — The sample size is 1 and therefore no standard deviation is available. | 2.1 (0.4) | 2.2 (0.5)
  4 Years: number analyzed (Participants) | 0 | 0 | 9 | 5
  4 Years |  |  | 2.1 (0.4) | 2.2 (0.4)
  5 Years: number analyzed (Participants) | 1 | 0 | 7 | 8
  5 Years | 4.4 (NA) — The sample size is 1 and therefore no standard deviation is available. |  | 2.3 (0.3) | 2.1 (0.5)

10. Secondary Outcome: Subject's Average Doppler Velocity Index (DVI)
Description: The Doppler Velocity Index (DVI) is a calculation of the ratio of the sub valvular velocity obtained by pulse wave Doppler and the maximum velocity obtained by continuous wave Doppler across the prosthetic valve, i.e. Time velocity interval (TVI) of the pulmonic valve / TVI of the RVOT. There are no normal ranges issued by the American Society of Echocardiography's Guidelines and Standards Committee for the pulmonary valve, however the expectation is that DVI should remain relatively steady over time but will generally decrease as the degree of stenosis (narrowing or constriction of the valve opening) worsens.
Time Frame: Baseline, 30 days, 3 months, and annually thereafter for up to 5 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 21 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 23 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 25 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 27 mm
Number analyzed (Participants) | 1 | 3 | 12 | 10
Ratio
  Baseline: number analyzed (Participants) | 0 | 2 | 5 | 6
  Baseline |  | 0.7 (0.1) | 0.6 (0.1) | 0.6 (0.2)
  30 days: number analyzed (Participants) | 0 | 0 | 8 | 6
  30 days |  |  | 0.5 (0.0) | 0.5 (0.1)
  3 months: number analyzed (Participants) | 1 | 1 | 10 | 5
  3 months | 0.7 (NA) — The sample size is 1 and therefore no standard deviation is available. | 0.5 (NA) — The sample size is 1 and therefore no standard deviation is available. | 0.5 (0.1) | 0.4 (0.1)
  1 Year: number analyzed (Participants) | 1 | 0 | 9 | 9
  1 Year | 0.5 (NA) — The sample size is 1 and therefore no standard deviation is available. |  | 0.4 (0.1) | 0.5 (0.1)
  2 Years: number analyzed (Participants) | 1 | 1 | 9 | 6
  2 Years | 0.5 (NA) — The sample size is 1 and therefore no standard deviation is available. | 0.4 (NA) — The sample size is 1 and therefore no standard deviation is available. | 0.5 (0.1) | 0.5 (0.1)
  3 Years: number analyzed (Participants) | 1 | 1 | 8 | 7
  3 Years | 0.3 (NA) — The sample size is 1 and therefore no standard deviation is available. | 0.4 (NA) — The sample size is 1 and therefore no standard deviation is available. | 0.5 (0.2) | 0.4 (0.1)
  4 Years: number analyzed (Participants) | 0 | 0 | 5 | 4
  4 Years |  |  | 0.4 (0.1) | 0.5 (0.2)
  5 Years: number analyzed (Participants) | 1 | 0 | 5 | 7
  5 Years | 0.2 (NA) — The sample size is 1 and therefore no standard deviation is available. |  | 0.4 (0.1) | 0.6 (0.1)

11. Secondary Outcome: Subject's Average Transvalvular Velocity Time Interval (VTI)
Description: Transvalvular regurgitation velocity time interval (VTI) is defined as the measurement in centimeters of the blood flowing backwards through the tricuspid valve, averaged over time. There are no defined normal ranges for VTI. The VTI value is dependent on the function of the right ventricle of the heart (chamber within the heart that is responsible for pumping oxygen-depleted blood to the lungs) and the expectation is the value should be relatively steady over time.
Time Frame: Baseline, 30 days, 3 months, and annually thereafter for up to 5 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 21 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 23 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 25 mm | Edwards Pericardial Aortic Bioprosthesis Model 11000A - 27 mm
Number analyzed (Participants) | 1 | 3 | 12 | 10
cm
  Baseline: number analyzed (Participants) | 0 | 2 | 8 | 5
  Baseline |  | 70.2 (7.3) | 82.9 (35.4) | 76.5 (12.0)
  30 days: number analyzed (Participants) | 0 | 0 | 7 | 6
  30 days |  |  | 77.8 (19.7) | 69.0 (17.2)
  3 Months: number analyzed (Participants) | 0 | 2 | 8 | 6
  3 Months |  | 73.9 (11.9) | 86.9 (16.8) | 75.9 (15.5)
  1 Year: number analyzed (Participants) | 1 | 1 | 8 | 8
  1 Year | 61.1 (NA) — The sample size is 1 and therefore no standard deviation is available. | 76.9 (NA) — The sample size is 1 and therefore no standard deviation is available. | 82.4 (18.8) | 73.9 (13.8)
  2 Years: number analyzed (Participants) | 0 | 1 | 8 | 7
  2 Years |  | 77.3 (NA) — The sample size is 1 and therefore no standard deviation is available. | 81.3 (17.2) | 64.1 (15.4)
  3 Years: number analyzed (Participants) | 0 | 1 | 8 | 7
  3 Years |  | 87.9 (NA) — The sample size is 1 and therefore no standard deviation is available. | 73.1 (18.5) | 70.3 (16.8)
  4 Years: number analyzed (Participants) | 0 | 0 | 7 | 5
  4 Years |  |  | 96.0 (16.9) | 79.1 (16.9)
  5 Years: number analyzed (Participants) | 0 | 1 | 6 | 7
  5 Years |  | 98.7 (NA) — The sample size is 1 and therefore no standard deviation is available. | 79.3 (20.3) | 74.1 (18.1)

12. Secondary Outcome: Change in Subject's New York Heart Association (NYHA)/Modified Ross Heart Failure Functional Class
Description: The New York Heart Association (NYHA)/Modified Ross functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, shortness of breath.
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath.
  Class III. Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or shortness of breath.
  Class IV. Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Changes in NYHA/Modified Ross HF classification from the preoperative baseline to the respective completed follow-up visits are shown as the number of subjects in each class who improved, worsened, or stayed the same.
Time Frame: Baseline, 30 days, 3 months, and annually thereafter for up to 5 years
Population: This outcome is reported for subjects who received the trial valve. Note that the number of participants analyzed is different from that in the participant flow as there was some missing data. NYHA was performed for subjects ≥13 years and the Modified Ross was performed for subjects ≤12 years. The following subjects converted to NYHA from Ross at the follow-up visit(s) due to meeting the age criteria: #6 at 5 Year, #7 at 5 Year, #13 at 4 Year and 5 Year, #22 at 3 Year, 4 Year and 5 Year.
Measure: Count of Participants; unit: Participants
Groups:
- Edwards Pericardial Aortic Bioprosthesis Model 11000A - Class I; Edwards Pericardial Aortic Bioprosthesis Model 11000A - Class II; Edwards Pericardial Aortic Bioprosthesis Model 11000A - Class III; Edwards Pericardial Aortic Bioprosthesis Model 11000A - Class IV: Edwards Pericardial Aortic Bioprosthesis Model 11000A in the pulmonary position in subjects five years or older requiring replacement of their native or prosthetic pulmonary valve.
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A - Class I | Edwards Pericardial Aortic Bioprosthesis Model 11000A - Class II | Edwards Pericardial Aortic Bioprosthesis Model 11000A - Class III | Edwards Pericardial Aortic Bioprosthesis Model 11000A - Class IV
Number analyzed (Participants) | 26 | 26 | 0 | 0
Participants
  30 days: number analyzed (Participants) | 16 | 10 | 0 | 0
  30 days: Improved | 0 | 10 | 0 | 0
  30 days: Same | 16 | 0 | 0 | 0
  30 days: Worsened | 0 | 0 | 0 | 0
  3 months: number analyzed (Participants) | 14 | 10 | 0 | 0
  3 months: Improved | 0 | 10 | 0 | 0
  3 months: Same | 14 | 0 | 0 | 0
  3 months: Worsened | 0 | 0 | 0 | 0
  1 year: number analyzed (Participants) | 15 | 10 | 0 | 0
  1 year: Improved | 0 | 10 | 0 | 0
  1 year: Same | 15 | 0 | 0 | 0
  1 year: Worsened | 0 | 0 | 0 | 0
  2 years: number analyzed (Participants) | 14 | 9 | 0 | 0
  2 years: Improved | 0 | 9 | 0 | 0
  2 years: Same | 14 | 0 | 0 | 0
  2 years: Worsened | 0 | 0 | 0 | 0
  3 years: number analyzed (Participants) | 15 | 9 | 0 | 0
  3 years: Improved | 0 | 9 | 0 | 0
  3 years: Same | 14 | 0 | 0 | 0
  3 years: Worsened | 1 | 0 | 0 | 0
  4 years: number analyzed (Participants) | 11 | 7 | 0 | 0
  4 years: Improved | 0 | 5 | 0 | 0
  4 years: Same | 9 | 2 | 0 | 0
  4 years: Worsened | 2 | 0 | 0 | 0
  5 years: number analyzed (Participants) | 14 | 8 | 0 | 0
  5 years: Improved | 0 | 8 | 0 | 0
  5 years: Same | 13 | 0 | 0 | 0
  5 years: Worsened | 1 | 0 | 0 | 0

13. Other Pre Specified Outcome: Subject's Average White Blood Cell Count
Description: Laboratory analysis of White Blood Cell (WBC) count on blood drawn from subject; WBC fight infection. The normal reference range for WBC count is 4.5 to 10.0 10^3 cells/microliters. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: Baseline, Discharge, 30 days, 3 months, and annually for up to 5 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliters
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 26
10^3 cells/microliters
  Baseline | 5.94 (1.41)
  Discharge | 7.40 (2.12)
  30 days: number analyzed (Participants) | 19
  30 days | 7.60 (2.47)
  3 months: number analyzed (Participants) | 17
  3 months | 6.15 (1.38)
  1 year: number analyzed (Participants) | 18
  1 year | 5.57 (1.24)
  2 years: number analyzed (Participants) | 13
  2 years | 6.13 (1.35)
  3 years: number analyzed (Participants) | 12
  3 years | 5.70 (1.74)
  4 years: number analyzed (Participants) | 8
  4 years | 6.02 (1.43)
  5 years: number analyzed (Participants) | 8
  5 years | 6.55 (1.02)

14. Other Pre Specified Outcome: Subject's Average Red Blood Cell Count
Description: The red blood cell (RBC) count is a test that measures the number of oxygen-carrying blood cells in your blood. The red blood cell count normal range for women is 4.2 to 5.4 10^6 cells/microliters and for men is 4.7 to 6.1 10^6 cells/microliters. A high red blood cell count may indicate that you have a condition that's preventing you from getting enough oxygen. A low RBC may be caused by an infection, or a medical condition related to anemia. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: Baseline, Discharge, 30 days, 3 months, and annually for up to 5 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliter
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 26
10^6 cells/microliter
  Baseline | 4.70 (0.33)
  Discharge | 3.69 (0.37)
  30 days: number analyzed (Participants) | 18
  30 days | 4.25 (0.31)
  3 months: number analyzed (Participants) | 17
  3 months | 4.69 (0.26)
  1 year: number analyzed (Participants) | 18
  1 year | 4.62 (0.38)
  2 years: number analyzed (Participants) | 12
  2 years | 4.75 (0.41)
  3 years: number analyzed (Participants) | 12
  3 years | 4.47 (0.26)
  4 years: number analyzed (Participants) | 8
  4 years | 4.49 (0.31)
  5 years: number analyzed (Participants) | 7
  5 years | 4.46 (0.43)

15. Other Pre Specified Outcome: Subject's Average Hemoglobin Count
Description: This is the laboratory analysis of Hemoglobin count on blood drawn from subjects. Hemoglobin is an oxygen-carrying protein in red blood cells. In males, a healthy hemoglobin level is between 13.2 and 16.6 g/dL. In females, a hemoglobin count of between 11.6 and 15 g/dL is considered normal and healthy. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: Baseline, Discharge, 30 days, 3 months, and annually for up to 5 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 26
g/dL
  Baseline | 13.61 (1.47)
  Discharge | 10.80 (1.07)
  30 days: number analyzed (Participants) | 19
  30 days | 12.18 (1.17)
  3 months: number analyzed (Participants) | 17
  3 months | 13.34 (1.04)
  1 year: number analyzed (Participants) | 18
  1 year | 13.62 (1.33)
  2 years: number analyzed (Participants) | 13
  2 years | 14.13 (1.41)
  3 years: number analyzed (Participants) | 12
  3 years | 13.06 (1.59)
  4 years: number analyzed (Participants) | 8
  4 years | 13.84 (0.89)
  5 years: number analyzed (Participants) | 8
  5 years | 13.11 (1.16)

16. Other Pre Specified Outcome: Subject's Average Hematocrit Percentage
Description: This is laboratory analysis of Hematocrit percentage on blood drawn from subjects. A hematocrit test measures the proportion of red blood cells in your blood. Red blood cells carry oxygen throughout your body. Having too few or too many red blood cells can be a sign of certain diseases. Normal hematocrit ranges for adult females are 36% to 44% and for adult males are 41% to 50%. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: Baseline, Discharge, 30 days, 3 months, and annually for up to 5 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 26
Percentage of red blood cells
  Baseline | 41.17 (3.51)
  Discharge | 32.35 (2.97)
  30 days: number analyzed (Participants) | 19
  30 days | 37.22 (3.30)
  3 months: number analyzed (Participants) | 17
  3 months | 40.47 (2.99)
  1 year: number analyzed (Participants) | 18
  1 year | 40.86 (3.53)
  2 years: number analyzed (Participants) | 13
  2 years | 41.88 (3.61)
  3 years: number analyzed (Participants) | 12
  3 years | 39.81 (4.05)
  4 years: number analyzed (Participants) | 8
  4 years | 41.61 (2.92)
  5 years: number analyzed (Participants) | 8
  5 years | 40.30 (3.90)

17. Other Pre Specified Outcome: Subject's Average Platelet Count
Description: This is laboratory analysis of Platelet count on blood drawn from subjects. The purpose of platelets is to create hemostasis, which is the prevention of hemorrhaging (bleeding) and the process of keeping blood inside the vessel walls. A normal platelet range is 150 to 450 10^3 cells/microliter. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: Baseline, Discharge, 30 days, 3 months, and annually for up to 5 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 26
10^3 cells/microliter
  Baseline | 223.04 (55.45)
  Discharge | 183.42 (54.00)
  30 days: number analyzed (Participants) | 19
  30 days | 304.84 (108.21)
  3 months: number analyzed (Participants) | 17
  3 months | 249.06 (70.77)
  1 year: number analyzed (Participants) | 18
  1 year | 240.17 (67.06)
  2 years: number analyzed (Participants) | 13
  2 years | 242.77 (64.46)
  3 years: number analyzed (Participants) | 12
  3 years | 252.17 (69.17)
  4 years: number analyzed (Participants) | 8
  4 years | 229.75 (89.74)
  5 years: number analyzed (Participants) | 8
  5 years | 232.25 (48.12)

18. Other Pre Specified Outcome: Subject's Average Serum LDH
Description: The lactate dehydrogenase (LDH) test looks for signs of damage to the body's tissues. Normal levels of LDH in the blood can vary depending on the lab, but usually range between 140 units per liter (U/L) to 280 U/L for adults and tend to be higher for children and teens.
Time Frame: Baseline, Discharge, 30 days, 3 months, and annually for up to 5 years
Population: This outcome is reported for subjects who received the trial valve. Note that the number of participants analyzed is different from that in the participant flow as there was some missing data. The protocol allowed subjects to have the option of having a serum LDH test or plasma free hemoglobin test or a haptoglobin test at each timeframe. Not all three tests were required for the subject.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 21
U/L
  Baseline: number analyzed (Participants) | 16
  Baseline | 153.69 (32.84)
  Discharge: number analyzed (Participants) | 17
  Discharge | 282.82 (61.92)
  30 days: number analyzed (Participants) | 13
  30 days | 207.77 (34.15)
  3 months: number analyzed (Participants) | 17
  3 months | 224.59 (49.81)
  1 year: number analyzed (Participants) | 17
  1 year | 201.00 (45.37)
  2 years: number analyzed (Participants) | 13
  2 years | 199.15 (40.50)
  3 years: number analyzed (Participants) | 10
  3 years | 209.50 (44.07)
  4 years: number analyzed (Participants) | 8
  4 years | 203.75 (37.16)
  5 years: number analyzed (Participants) | 5
  5 years | 192.60 (22.81)

19. Other Pre Specified Outcome: Subject's Average Plasma Free Hemoglobin
Description: Laboratory Analysis of Plasma Free Hemoglobin (Hgb) of blood drawn from subject. This blood test measures the level of free hemoglobin in the plasma (liquid portion of the blood). The reference range for plasma free hemoglobin is 0.0 to 15.2 mg/dL. In general, values higher than this can indicate something is wrong.
Time Frame: Baseline, Discharge, 30 days, 3 months, and annually for up to 5 years
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 5
mg/dl
  Baseline | 45.00 (33.54)
  Discharge: number analyzed (Participants) | 1
  Discharge | 30.00 (NA) — The sample is 1 and therefore no standard deviation is available.
  30 days: number analyzed (Participants) | 0
  3 months: number analyzed (Participants) | 0
  1 year: number analyzed (Participants) | 1
  1 year | 5.80 (NA) — The sample is 1 and therefore no standard deviation is available.
  2 years: number analyzed (Participants) | 0
  3 years: number analyzed (Participants) | 0
  4 years: number analyzed (Participants) | 0
  5 years: number analyzed (Participants) | 0

20. Other Pre Specified Outcome: Subject's Average International Normalized Ratio (INR)
Description: The INR is a calculation based on results of a prothrombin time (PT). The PT is a blood test that measures the time it takes for the liquid portion (plasma) of the blood to clot. The normal range of INR depends on the patient. If they are not on an anticoagulant therapy, then the normal range is 0.9 - 1.1 and if they are on anticoagulant therapy then the normal range is 2 - 3.
Time Frame: Baseline, Discharge, 30 days, 3 months, and annually for up to 5 years
Population: This outcome is reported for subjects who received the trial valve who were on anticoagulant therapy during the trial. Note that only three of the 26 total participants were on anticoagulant therapy and that the number of participants analyzed is different from that in the participant flow as there was also some missing data.
Measure: Mean (Standard Deviation); unit: Ratio of blood clotting
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 3
Ratio of blood clotting
  Baseline | 1.05 (0.02)
  Discharge: number analyzed (Participants) | 2
  Discharge | 1.23 (0.27)
  30 days: number analyzed (Participants) | 1
  30 days | 1.99 (NA) — The sample size is 1 and therefore no standard deviation is available.
  3 months: number analyzed (Participants) | 0
  1 year: number analyzed (Participants) | 1
  1 year | 2.45 (NA) — The sample size is 1 and therefore no standard deviation is available.
  2 years: number analyzed (Participants) | 0
  3 years: number analyzed (Participants) | 1
  3 years | 1.02 (NA) — The sample size is 1 and therefore no standard deviation is available.
  4 years: number analyzed (Participants) | 0
  5 years: number analyzed (Participants) | 0

21. Other Pre Specified Outcome: Subject's Average Urine Urobilinogen (if Necessary for Subjects 12 Years and Under)
Description: Urobilinogen is a substance that is produced when bilirubin, a waste product produced by the breakdown of red blood cells, is processed in the liver and released into the intestine. The normal range of urobilinogen is less than 1 mg/dL. It is common to have values within the 0 to 8 mg/dL range. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: Baseline, Discharge, 30 days, 3 months, and annually for up to 5 years
Population: This outcome is reported for subjects who received the trial valve and required the urine urobilinogen clinical test. There were no subjects in the trial who required this clinical test.
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through five years post-implant.
Description: The outcome is site reported for subjects who received the Edwards Pericardial Aortic Bioprosthesis Model 11000A device in the pulmonary position where data is available.
Arm/Group | Edwards Pericardial Aortic Bioprosthesis Model 11000A
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 10/26
Other Adverse Events (participants affected / at risk) | 22/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards Pericardial Aortic Bioprosthesis Model 11000A (N=26)
NONSPECIFIC, UNKNOWN, OR OTHER BODY SYSTEM | ALLERGIC REACTION - MEDICATION RELATED (General disorders) | 1 (1)
NONSPECIFIC, UNKNOWN, OR OTHER BODY SYSTEM | ANAPHYLACTIC REACTION (General disorders) | 1 (1)
CARDIOVASCULAR - ARRHYTHMIA | ARRHYTHMIA - ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
CARDIOVASCULAR - ARRHYTHMIA | ARRHYTHMIA - TACHYCARDIA -VENTRICULAR (Cardiac disorders) | 1 (1)
BLOOD AND LYMPHATIC (INCLUDING ALL BLEEDING COMPLICATIONS) | BLEEDING - CARDIOVASCULAR - MAJOR (Blood and lymphatic system disorders) | 1 (1)
BLOOD AND LYMPHATIC (INCLUDING ALL BLEEDING COMPLICATIONS) | BLEEDING - GASTROINTESTINAL UPPER - MAJ (Blood and lymphatic system disorders) | 1 (1)
CARDIOVASCULAR - MISC | PERICARDIAL EFFUSION - MINOR (Cardiac disorders) | 1 (1)
MUSCULAR SKELETAL/DERMATOLOGIC | STERNAL WOUND/THORACIC INFECTION (Musculoskeletal and connective tissue disorders) | 1 (1)
CARDIOVASCULAR - ARRHYTHMIA | ARRHYTHMIA - SUPRAVENTRICULAR TACHYCARDIA (SVT) (Cardiac disorders) | 1 (1)
CARDIOVASCULAR - REGURGITATION | REGURGITATION - PULMONARY-CENTRAL/TRANSVALVULAR-+3 (Cardiac disorders) | 2 (2)
CARDIOVASCULAR - REGURGITATION | REGURGITATION - PULMONARY-CENTRAL/TRANSVALVULAR-+4 (Cardiac disorders) | 1 (1)
CARDIOVASCULAR - STENOSIS | STENOSIS - PULMONARY - MODERATE (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards Pericardial Aortic Bioprosthesis Model 11000A (N=26)
CARDIOVASCULAR - ARRHYTHMIA | ARRHYTHMIA - AV BLOCK - 1ST DEGREE (Cardiac disorders) | 2 (2)
CARDIOVASCULAR - ARRHYTHMIA | ARRHYTHMIA - OTHER (Cardiac disorders) | 2 (2)
CARDIOVASCULAR - MISC | CARDIOVASCULAR - OTHER (Cardiac disorders) | 2 (2)
CARDIOVASCULAR - REGURGITATION | REGURGITATION - PULMONARY-CENTRAL/TRANSVALVULAR-+3 (Cardiac disorders) | 10 (10)
CARDIOVASCULAR - REGURGITATION | REGURGITATION - PULMONARY-CENTRAL/TRANSVALVULAR-+4 (Cardiac disorders) | 4 (4)
CARDIOVASCULAR - STENOSIS | STENOSIS - PULMONARY - MODERATE (Cardiac disorders) | 2 (2)
MUSCULAR SKELETAL/DERMATOLOGIC | MUSCULAR SKELETAL / DERMATOLOGIC - OTHER (Musculoskeletal and connective tissue disorders) | 2 (3)
NONSPECIFIC, UNKNOWN, OR OTHER BODY SYSTEM | NONSPECIFIC, UNKNOWN OR OTHER BODY SYSTEM - OTHER COMPL (General disorders) | 4 (5)
PULMONARY/RESPIRATORY | ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 8 (8)
PULMONARY/RESPIRATORY | PLEURAL EFFUSION - BILATERAL (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can't publish/present on overall study results not yet published but may publish his own data subject to EW review. Manuscripts will be submitted to EW for review 30 days prior to submission of manuscript for publication/presentation. EW may ask for a 60 day delay to protect proprietary information/filing of related patent applications. Site-specific results of devices which haven't been market released shall not include claims of device safety/effectiveness and require EW review/approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT02656290/Prot_SAP_000.pdf